CLINICAL TRIAL: NCT07099755
Title: Effect of Dynamic Neuro-musclar Stabilization on Woman With Post Partum Low Back Pain
Brief Title: This Study Aimed to Evaluate the Effect of Dynamic Neuromuscular Stabilization (DNS) on Pain Intensity and Functional Disability in Women With PLBP as Common Problem Affect t he Women After Birth Which Often Impacting Their Quality of Life and Ability to Perform Daily Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gehad Alaa (Other)
Responsible Party: Sponsor-Investigator, Gehad Alaa, Gehad alaa mohy el-deen abd el-raheem, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: No:P.T.REC/012/005604
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-07

CONDITIONS: Post -Partum Low Back Pain; Dynamic Neuromuscular Stabilization (DNS); Women's Health / Physiotherapy; Musculoskeletal Rehabilitation; Core Stability and Functional Disability
MeSH Terms: interventions — Exercise; Ultrasonography

STUDY DESIGN:
Intervention Model Description: This study employed a parallel assignment interventional model in which 60 postpartum women with low back pain were randomly assigned to one of two groups:
  Experimental Group: Received Dynamic Neuromuscular Stabilization (DNS) exercises in addition to conventional therapy (ultrasound and infrared therapy).
  Control Group: Received only conventional therapy without DNS.
  Both groups followed the assigned intervention protocol 3 times per week for 6 weeks. Outcome measures (pain intensity and functional disability) were assessed at baseline and after the intervention period using the Numeric Pain Rating Scale (NPRS) and Modified Oswestry Disability Questionnaire (MODQ).
  Randomization ensured comparable baseline characteristics and minimized selection bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arms (Experimental): Intervention Group (Experimental Arm):
  Participants in this group received a comprehensive physiotherapy program consisting of:
  Ultrasound therapy (continuous mode, 1 MHz, 1.5 W/cm² for 5 minutes),
  Infrared therapy (15 minutes per session),
  Dynamic Neuromuscular Stabilization (DNS) exercises focused on breathing control, core activation, and developmental movement patterns (e.g., supine 90/90, quadruped, side-lying, etc.), administered 3 times per week for 6 weeks.
  Interventions: Behavioral: Intervention Group: Name: Dynamic Neuromuscular Stabilization (DNS) Exercises
- Control Group (Conventional Treatment Arm): (Experimental): Participants in this group received the same physiotherapy program as the intervention group Ultrasound therapy (continuous mode, 1 MHz, 1.5 W/cm² for 5 minutes) Infrared therapy (15 minutes per session), but without DNS exercises.
  Interventions: Device: Control Group:Name: Conventional Physiotherapy (Ultrasound and Infrared Therapy)

INTERVENTIONS:
Behavioral: Intervention Group: Name: Dynamic Neuromuscular Stabilization (DNS) Exercises — Distinguishing Description for DNS Intervention
  This intervention consists of a structured Dynamic Neuromuscular Stabilization (DNS) exercise program specifically tailored for post-partum women with mechanical low back pain. DNS emphasizes restoring functional motor patterns through:
  Breathing-based core activation techniques
  Developmental positions mimicking infant motor milestones (e.g., supine 90/90, quadruped, side-lying)
  Coordination of the diaphragm, pelvic floor, and transverse abdominis muscles
  Progressive motor control retraining over 6 weeks, 3 sessions/week
  What distinguishes this intervention:
  It integrates developmental kinesiology principles with respiratory-pelvic-lumbar coordination.
  DNS is performed under supervised sessions by a physiotherapist, ensuring precision and progression.
  This protocol replaces standard strengthening/stretching exercises and focuses on neuromuscular re-patterning, not just symptom relief.
  Other Names: Behavioral Physiotherapy for PLBP; Postural Motor Control Exercises; Core Stabilization Exercises; DNS Training
  Arms: Study Arms
Device: Control Group:Name: Conventional Physiotherapy (Ultrasound and Infrared Therapy) — 1-Therapeutic Ultrasonic: comparison group also received treatment through therapeutic ultrasound, which was applied three times per week. The ultrasound therapy was delivered to the paraspinal muscles of the lumbar region, using a stroking technique where each stroke overlapped by about 50% with the preceding stroke. The ultrasound used a frequency of 3 MHz and an intensity range of 1.0 to 1.5 W/cm²,The ultrasound head was placed over the L4 to L5 and L5 to S1 regions and moved in a circular motion for a total duration of 5 minutes per treatment session (Shobari et al., 2024).
  infra red the infrared lamp was placed at 75 cm distance from the patient's back so that the radiation struck the surface at or near a right angle to achieve maximum penetration. The treatment duration was 15 minutes. Each woman with post-partum low back pain was treated by 20 minutes infrared irradiation 40 cm away from the low back region, from prone3 sessions per week for 6 weeks (El-Lassy and Madian, 2018
  Other Names: Standard Physical Therapy; US + IR Therapy; Non-exercise-based conservative treatment; Control group treatment protocol
  Arms: Control Group (Conventional Treatment Arm):

SUMMARY:
The aim of this study was to determine the effect of DNS on women with post-partum LBP.

Post-partum low back pain (PLBP) represents a prevalent and clinically significant condition that adversely impacts mobility, pelvic floor integrity, functional performance, and quality of life in women following childbirth. Epidemiological data suggest that approximately 50% of women who experience pregnancy-related low back pain continue to report symptoms up to 12 months post-partum, while nearly 20% may develop chronic or disabling pain lasting up to three years. Moreover, the onset of LBP within the first three months postpartum is a strong predictor for the development of persistent or recurrent symptoms, emphasizing the importance of early intervention (Fukano et al., 2021).

Dynamic Neuromuscular Stabilization (DNS) provides a novel and integrative rehabilitation framework based on developmental kinesiology, emphasizing the restoration of optimal joint centration, intra-abdominal pressure regulation, and neuromuscular coordination across the entire core system. DNS targets not just local symptoms but the underlying movement dysfunctions that contribute to persistent post-partum pain. This approach stands in contrast to traditional rehabilitation techniques that often emphasize symptomatic relief over functional re-patterning (Ghavipanje et al., 2021).

The significance of this study lies in its investigation of DNS as an evidence-based, functional intervention for women with PLBP. It highlights the role of active patient engagement, corrective movement strategies, and motor control retraining in promoting long-term recovery. By demonstrating the effectiveness of DNS, this research contributes to the evolving body of literature supporting core-centric, integrated neuromuscular rehabilitation for post-partum populations, with potential implications for improving clinical outcomes and enhancing women's physical autonomy after childbirth.

Delimitations

The present study was delimited to the following criteria to ensure homogeneity of the sample and clinical relevance to post-partum rehabilitation:

1. Participants: Sixty post-partum women diagnosed with mechanical low back pain of 3 to 6 months duration were included, reflecting a subacute pain profile relevant for neuromuscular retraining.
2. Age Range: Participants were between 18 and 34 years of age, corresponding to typical reproductive and early post-partum demographic profiles.
3. Body Mass Index (BMI): Only individuals with a BMI between 25 kg/m² and 35 kg/m² were included to account for mild to moderate overweight status, a known factor in post-partum back dysfunction.
4. Medication Exclusion: Participants did not receive any analgesics, anti-inflammatories, or therapeutic interventions throughout the study period to eliminate confounding effects.
5. Medical Exclusion: Women with a history of severe trauma, skeletal injuries, fractures, neurologic or chronic inflammatory disorders, primary or metastatic neoplasms, osteoporosis, or chronic neuromuscular conditions contributing to LBP were excluded.
6. Consent and Stability: Only medically stable women who provided written informed consent were included, in line with ethical standards for human subject research.

Limitations

Despite careful design and standardized intervention protocols, the current study was subject to several limitations inherent in clinical research involving post-partum populations:

1. Emotional and Psychological Factors: The emotional state of post-partum women - including symptoms of fatigue, anxiety, or depressive mood - may have influenced motivation, engagement, and consistency during therapeutic sessions. These psychosocial elements are known to modulate both pain perception and motor performance (Morin et al., 2018).
2. Participant Cooperation and Compliance: Variability in the degree of cooperation and adherence to prescribed home exercises may have introduced inconsistencies in treatment effects. Factors such as childcare responsibilities and sleep disturbances can influence session attendance and follow-through (Boissonnault & Blanpied, 2018).
3. Individual Response to Therapy: There may have been biological and neuromuscular differences in how participants responded to the DNS approach. Genetic variability, post-partum recovery rate, and prior physical activity levels are all variables that can modulate treatment outcomes (Kolar et al., 2014).
4. Motor Learning and Skill Acquisition: DNS-based exercises require a level of motor learning and sensory awareness, which varies among individuals. Differences in performance ability and learning curve may have affected the precision and efficiency with which patients executed the exercises (Kolar et al., 2012).
5. Socioeconomic and Cultural Differences: Economic status, educational background, and cultural norms influenced participants' access to resources, health beliefs, and commitment to therapeutic regimens. (smith et al.2023)

DETAILED DESCRIPTION:
I- Design of Study:

The study was designed as a randomized, pre-post-test study. Setting This study was conducted at the Outpatient Physical Therapy Clinic of Saqulta Central Hospital, Sohag, Egypt, and aimed to examine the therapeutic impact of Dynamic Neuromuscular Stabilization (DNS) on pain intensity and functional disability in women suffering from post-partum low back pain (LBP). DNS, as a clinical application of neurodevelopmental kinesiology, utilizes developmental postures and breathing coordination to re-establish intrinsic trunk stability.

The duration of the study extended from the forth of December 2024 to fifth of May 2025, during which participants underwent DNS-based intervention under standardized clinical protocols. The environment was controlled to ensure consistency in therapeutic delivery and outcome measurement, aligning with similar methodological approaches in neuromuscular rehabilitation research (Kolar et al., 2012).

III- Subjects' criteria:

The study recruited 60 postpartum women experiencing low back pain (LBP) from the outpatient clinic of Saqulta Central Hospital, Sohag, Egypt. Participants with post-partum low back pain aged 18-34 years, with a BMI of 25-35 kg/m², and reported LBP intensity ≥5 on the Numeric Rating Scale (NRS), localized between T12 and the gluteal folds (with possible lower extremity involvement). All participants had a disability score ≥20% on the Modified Oswestry Disability Questionnaire (MODQ). Women were excluded if they had gynecological conditions (e.g., endometriosis, ovarian cysts, uterine fibroids), orthopedic/spinal disorders (e.g., trauma, scoliosis, pre-existing non-postpartum LBP), or systemic pathologies (e.g., inflammatory diseases, malignancy, osteoporosis, neurological deficits). Additional exclusions included recent fractures, chronic neuromuscular disorders, or concurrent analgesic use during the study.

IV- Ethical approval The evaluation and treatment protocol were explained to each patient. A detailed evaluation sheet was made for each patient. A brief explanation was given to the patient of the assessment procedures for each patient. Each patient signed a consent form prior to conducting the study. The protocol was approved by the Ethical Committee of the Faculty of Physiotherapy, Cairo University with number: (No: P.T.REC/012/005604 on 3/12/2024).

V- Sampling and randomization The sample size calculation was done by G-Power 3.1.9.2 (Universitat Kiel, Germany). The mean ± SD of Numeric Pain Rating Scale (NPRS) was 5.06 ± 1.09 in group A and was 4.29 ± 0.92 in group B according to a previous study (Park et al., 2021). The sample size was based on the following considerations: 0.763 effect size, 95% confidence limit, 80% power of the study, group ratio 1:1 and two cases were added to each group to overcome dropout. Therefore, we recruited 30 patients in each group.

Patients were randomized into two equal groups in a parallel manner by computer generated numbers and their allocation code was kept in a closed opaque envelope:

* Group A (Control Group) (n=30): Women was treated by ultrasonic therapy and infrared, 3 sessions per week for 6 weeks.
* Group B (Study Group) (n=30): Women was treated by ultrasonic therapy, infrared and dynamic neuro- muscular stabilization.

This study was open label. 79 patients were assessed for eligibility, 13 patients did not meet the criteria, and 6 patients refused to participate in the study. The remaining patients were randomly allocated into two equal groups (30 patients in each). All allocated patients were followed up and analyzed statistically flowchart (Figure 18).

Every patient had a secret code number. All data of the patients were confidential with secret codes and private files for each patient; all given data was used for the current medical research only.

All participants were given a full explanation of the study protocol, and a consent form was signed by each patient before entry into the study.

VI- Instrumentation

The main equipment and tools are classified into two main categories:

A. Evaluative instrumentations:

1. Recording datasheet:

   Demographic data: all information of each female in this study including name, age, address, occupation, weight, height, body mass index (BMI), number of parity and gravity, gestational age (assessment from the date of the last menstrual period), present history, medical history, past history and family history to confirm that there were no contraindications that interfere with the study and all measuring variables were collected on the recording data sheet .
2. Weight and height scale: It was used to measure the body weight and height of each woman in both groups (A and B) before the beginning of the study to calculate BMI according to formula: BMI (kg/m2) = weight /height2 before the starting of treatment procedures .
3. Numeric pain-rating scale (NPRS):

   NPRS was applied to assess the severity of pain for both groups A and B pre and post the intervention. The NPRS extends from 0 (no pain) to 10 (very severe pain) and showed adequate and high test-retest reliability. The participants circled the numerical value on the segmented scale to indicate pain level, its simplicity, reliability, and validity as well as its ratio scale properties make the NPRS the optional tool for describing pain intensity.
4. Modified Oswestry Disability Questionnaire (MODQ):

MODQ was used to assess pain-related disability for each woman in both groups (A&B), the secondary outcome involved the impact of LBP on daily activities. MODQ as a functional scale assesses the effects of LBP on daily activities by assigning a disability score daily activities (disability score) and the respondent's fear avoidance beliefs about LBP. The MODQ as a functional scale assesses the effects of LBP on daily activities by assigning a disability score, according to the answered question according to the answered questions The MODQ contains 10 questions regarding the level of pain and interference with several daily physical activity including sleeping, self-care, lifting, traveling, and social life every question is scored on a 6-point scale (0-5), and participants are requested to option, The Arabic version of the Oswestry Disability Index is a highly valid tool for assessing self-reported disability in patients with low back pain and demonstrates excellent test-retest reliability .

B. Treatment instrumentation:

1. Therapeutic Ultrasonic:

   Ultrasonic device Phyaction 190i, Uniphy P.O. Box 558, serial number 2745, End hoven, The Netherlands 230 V. Continuous Ultrasonic was applied for 5 minutes duration with 1W/cm2 intensity, frequency 1 MHz and 100% duty cycle. (Saleh et al., 2019; Haile et al., 2021) .
2. Infrared device :

4004/2N, Verreet Quartz Dixwell, France. The device has a power of 400 w, voltage 220 V and a frequency of 50/60 Hz . The infrared lamp was placed at 75cm distance from the patient's back so that the radiation struck the surface at or near a right angle to achieve maximum penetration. The treatment duration was 15 minutes, it was applied for groups, at frequency of 3 sessions per week for 6 weeks (Araujo et al., 2021, Saleh et al., 2019).

VII- Procedures A. Evaluative procedures:All patients were given a full explanation of the protocol of the study and a consent form was signed by each patient before participation in the study.

At baseline, all participants provided a medical history, underwent a standardized examination by a specialist in obstetrics and infertility as well as a physical therapy assessment, and completed a series of self-report questionnaires.

1. History Taking:

   A detailed medical history was taken from each woman before entry into the study and recorded in a recording data sheet.
2. Weight and height measurements:

   They were measured using Weight- height scale, for each participating woman in both groups (A and B) before starting the treatment via standing on the scale with light clothes and bare feet to calculate the BMI according to the following equation: BMI=Weight/Height2 (Kg/M2).
3. Pain Assessment:

   Pain intensity was assessed using the Numeric Pain Rating Scale (NPRS) for all participants in both groups, before and after the treatment program. Each woman marked a point on the scale corresponding to her pain intensity, with a 2-point change considered clinically meaningful and beyond measurement error. In this study, the NPRS demonstrated high test-retest reliability.
4. Disability assessment:

The Modified Oswestry Disability Questionnaire (MODQ) was done for all participating woman before and after the treatment.

MODQ is a standardized tool used to assess a patient's level of disability due to low back pain. It helps to measure the impact of back pain on a person's daily life and provides insights into the severity of the condition.

The questionnaire consists of 10 sections, each focusing on a different aspect of daily functioning, such as pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and sex life. Each section has a set of statements, and the patient must select the one that best represents their condition.

Each section was scored on a scale from 0 to 5, and the total score was calculated by summing the individual responses. The overall score was expressed as a percentage, with higher scores indicating greater disability.

The minimum clinically significant difference (MCID) for the MODQ has been reported as 6 points. Moreover, the Persian version of the MODQ is introduced as a valid and reliable tool for evaluating the disability following low back pain.

B. Treatment procedures:

1. Therapeutic Ultrasonic:

   In the current study, women suffering from post-partum low back pain were administered a therapeutic intervention using dynamic neuro-muscular stabilization (DNS) techniques. However, a comparison group also received treatment through therapeutic ultrasound, which was applied three times per week. The ultrasound therapy was delivered to the paraspinal muscles of the lumbar region, using a stroking technique where each stroke overlapped by about 50% with the preceding stroke. The ultrasound used a frequency of 3 MHz and an intensity range of 1.0 to 1.5 W/cm², applied in pulsed mode. The women were positioned comfortably in the prone position, with coupling gel applied to the skin over the treated area. The ultrasound head was placed over the L4 to L5 and L5 to S1 regions and moved in a circular motion for a total duration of 5 minutes per treatment session (Shobari et al., 2024).
2. Infrared device:

Both groups, each woman with post-partum low back pain was treated by the infrared lamp was placed at 75 cm distance from the patient's back so that the radiation struck the surface at or near a right angle to achieve maximum penetration. The treatment duration was 15 minutes. Each woman with post-partum low back pain was treated by 20 minutes infrared irradiation 40 cm away from the low back region, from prone position, 3 sessions per week for 6 weeks (El-Lassy and Madian, 2018).

3-DNS exercise program: The intervention was applied only to Group B, conducted daily over a period of six weeks. Based on the Dynamic Neuromuscular Stabilization (DNS) approach, the exercise program included diaphragmatic breathing and a progression of postural positions: Baby Rock (supine 90-90), prone, rolling, side-lying, oblique sitting, tripod, kneeling, squat, and standing positions (Mahdieh et al., 2020a).

Each participant followed the DNS protocol, consisting of three supervised sessions and three home-based sessions per week throughout the six-week period. The exercises were first demonstrated using verbal instructions and visual aids, such as photographs, to ensure proper technique and understanding.

C. Methodology:

Expand the lower ribcage and abdominal wall proportionally during inhalation, Maintain balanced tension across the abdominal wall during exhalation, Adjust the pelvis, spine, ribcage, and scapulae into optimal alignment with manual/verbal cues from the therapist.

The exercises followed developmental kinesiology principles, progressing only upon mastery of prior movement patterns. Intensity was graded based on developmental positions (e.g., supine → quadruped → standing) to reinforce automatic stabilization and breathing synergies.

During the exercises, special attention was given to the breathing pattern, with emphasis on the stereotyped coordination of inhalation and exhalation. Participants were encouraged to expand the lower chest cavity and the entire abdominal wall proportionally during inhalation, and to maintain balanced tension across all abdominal wall sections during exhalation, as described in the DNS manual (Canales et al., 2017, Davidek et al., 2018, Mahdieh et al., 2020, Mohammad Rahimi et al., 2020).

The therapist provided both verbal and manual guidance to help participants achieve optimal alignment of the pelvis, spine, ribcage, and scapulae, while ensuring proper core stabilization across various developmental positions. Because the effectiveness of DNS depends on precise execution of postural and breathing patterns, the therapist closely supervised all stages of the exercise sessions.

Exercise intensity in the DNS group was determined according to the developmental positions outlined in DNS principles, which are based on the automatic activation patterns of postural-locomotor function and breathing derived from developmental kinesiology.

Supervised exercises were conducted three times a week (Saturday, Monday, and Wednesday), while home-based exercises were performed on Sunday, Tuesday, and Thursday. The home exercise program mirrored the supervised sessions in both number of exercises and repetitions. Prior to each home-based session, participants attended a supervised practice session to learn the correct technique and mechanics. To enhance accuracy and adherence, each participant received a booklet containing illustrated instructions for all exercises.

1. Week 1 (session duration 30 min daily) from following position:

   * Supine breathing exercise Participants were instructed to follow a specific breathing exercise protocol aimed at enhancing core stability and alleviating low back pain. For the first week of the program, participants performed the exercise daily, with each session lasting for 30 minutes. The exercise was done from a supine position, following a diaphragmatic breathing pattern: 10 repetitions, with a 1-second inhale and a 2-second exhale, followed by a 60-90 second rest in between each repetition . The breathing exercise aimed to promote core activation and was designed to improve overall stability for postpartum women suffering from low back pain (Mahdieh et al., 2020)..
   * Prone breathing exercise:

   Description: Participants performed a prone breathing exercise as part of their rehabilitation program. The exercise was carried out with the participants in a prone position, ensuring that the spine was kept in an upright position to maintain pelvic neutrality and avoid hyperextension of the cervical spine. This posture aimed to promote balanced activation of the scapula fixators. During the exercise, participants followed a diaphragmatic breathing pattern, performing 10 repetitions with a 1-second inhale and a 2-second exhale, followed by a 60-90 second rest between each repetition . The objective was to enhance core muscle activation and improve overall stability, contributing to the relief of postpartum low back pain (Mahdieh et al., 2020).

   • Breathing Exercise 90-90 Description: Supine by positioning face up and back on the floor with the feet on a wall, so the knees are bent to 90 degrees and the hips are bent to 90 degrees. The neck and spine should be "neutral" and comfortable. One hand on the upper chest and one hand on the lower abdomen, follow a diaphragmatic breathing pattern:10 repetitions with 1sec inhale, 2-sec exhalation, and 60-90 sec rest period .

   • Prone Position Elbow Support 90-90: Description: From prone position with elbow 90-90, weight-bearing on the medial epicondyles with the neck extension initiated in the mid thoracic segments (T3/4/5), the cervical and upper thoracic spine are maintained upright, with ideal alignment between the chest and the pelvis.

   Ordered to keep the pelvis in neutral and avoid hyperextension in the cervical spine and follow a manner of diaphragmatic breathing pattern: 10 repetitions with 1sec inhale and 2 sec exhale and 60-90 sec rest period ..
2. Week 2 (session duration 35 min) from the following position (Kong et al., 2024):

   • Supine Position 90-90-degree hip and knee flexion Arm Outside the Body (4-month-old position): Description: 90-degree hip flexion, functional centration at the hips, spine upright, shoulder girdles relaxed, chest and pelvis properly aligned (chest and pelvic axis parallel (Kong et al., 2024).

   From the position follows a diaphragmatic breathing pattern:10 repetitions with 1sec inhale ,2 sec exhale and 60-90 sec rest period .
   * Supine Position 90-90-degree hip and knee flexion Arm on The Abdomen (4-month-old position) Describtion: 90-degree hip flexion, functional centration at the hips, spine upright, shoulder girdles relaxed, chest and pelvis properly aligned (chest and pelvic axis parallel, From the position , follow a manner of diaphragmatic breathing pattern: 10 repetitions with 1sec inhale, 2 sec exhale and 60-90 sec rest period .
   * Creeping position (one hip and knee flexion), elbow support on ASIS. and medial epicondyle of the opposite knee (4.5-month position).

   Discribtion; Basic supine exercise, the hips are well-centrated during the entire exercise 90° flexion and slight external rotation at the hips. Support or weight bearing was at the level of the upper gluteal muscles.

   Precaution : the exercise should be discontinued if the back arches into extension or if the subject was unable to maintain the hip and knee position. From the posion, follow a manner of diaphragmatic breathing: 10 repetitions with 1sec inhale 2 sec and exhale and 60-90 sec rest period .
3. Week 3 (session duration 40min) from following positions (Kong et al., 2024):

   • Rolling pattern (ipsilateral position) Description: From side position with the upper and lower limbs in reciprocal differentiated function with the bottom extremities being activated in support function (closed kinetic chain) and top extremities in reaching/stepping forward function (closed kinetic chain).

   Keep spine and the pelvis in neutral position, follow a manner of diaphragmatic breathing pattern: 15 repetitions with 2 sec inhale, 4 sec. exhale with 60-90 sec rest period(Kong et al., 2024)
   * Supine Position 90-90-degree hip and knee flexion Hand on The Knee Description: Supine 90-90 hands on the knee Maintain the spine elongated and the pelvis in neutral, from this position, follow a manner of diaphragmatic breathing pattern: 15 repetitions with -2 sec inhale, 4 sec exhale with 60-90 sec rest period (Kong et al., 2024)
   * Prone Position Hand and Knee Support (elbow in an extension) (6-month-old position) Description: prone position with support on both medial epicondyles and the pubic symphysis with guiding the patient's shoulder blades to a neutral caudal position and neck extended focusing on initiating the movement at the mid-thoracic spinal segments and C7/T1/T2/T3/T4/T5.

   Take deep diaphragmatic inspiration and expand the latero-dorsal abdominal section maintaining the neutral chest position aiming to help the shoulder alignment and elongate the spine. Diaphragmatic Breathing manner: 15 repetitions with -2sec inhale 4 sec and exhale and 60-90 sec rest period .

   • Supine position hand on foot (4-month-old position) Description: Supine position, hip and knee 45-degree flexion, each hand on each foot on the same side. From this position, follow a breathing pattern aiming to help the shoulder alignment and elongate the spine manner of diaphragmatic breathing: 15 repetitions with 2sec inhale, 4 sec exhale with 60-90 sec rest period
4. Week 4 positions (session duration 45min) from following positions (4-month-old position):

   • Quadruped position: Description: quadruped with shift forward i.e the angle between the trunk and the hip 120 degree, from this position, follow breathing pattern aiming to help the shoulder alignment and elongate the spine.

   Diaphragmatic Breathing manner: 15 repetitions with -2sec inhale, 4 sec exhale and 60-90 sec rest period .

   • Quadruped position (the angle between the trunk and the hip 90 degree): Description: quadruped position with body segments properly aligned in which the shoulder girdles are positioned over the well-supported hands in a fully loaded neutral/concentrated position: weight distribution must be proportional on all metacarpophalangeal joints (equally on the thenar and hypothenar areas), the hip joints are in slight external rotation, positioned above the supported knees, while the shins and feet converge. The entire spine and the trunk are upright.

   From this position, follow breathing pattern aiming to help the shoulder alignment and elongate the spine. Diaphragmatic breathing manner: 15 repetitions with 2 sec inhale, 4 sec, exhale with 60-90 sec rest period .

   • Oblique and Siting Position (Side Plank) with Arm and Lateral Knee Support Description: Initial oblique side sitting position with the top leg supported on the floor, then Trunk rotation with arm reaching forward, lifting the pelvis in a side sitting position support shifting weight from the buttock toward the lateral condyle of the knee of the bottom leg, insuring the lower (supporting) scapula in caudal position adhering to the rib cage, its medial border parallel with the spine (not elevated or winging) then be stable. From this position, follow aiming to help the shoulder alignment and elongate the spine. Diaphragmatic Breathing manner: -15 repetitions with 2sec inhale, 4 sec exhales with 60-90 sec rest period.

   • An Oblique Siting Position with Hand Support (Elbow Extended) Description: Side Oblique sitting position with hand support by lifting the pelvis and loading the bottom knee, shoulder girdle stabilized neutral i.e. should not be winged.

   From this position, follow a breathing pattern aiming to help the shoulder alignment and elongate the spine. Diaphragmatic breathing manner:15 repetitions with 2sec inhale ,4 sec exhale with 60-90 sec rest period .

   • Crawling position (9-month position): Description: Training core stabilization while supported on all fours. Instruct the patient to elongate the spine, tuck the chin, and weight-bear on concentrated hands (proportional loading on the hands) and both knees.

   Exercise progression: Ask the patient to lift one arm then the contralateral leg and hold the position while correct joint centration and core stabilization are maintained. From this position, follow a manner of diaphragmatic breathing:15 hyperventilation with -2sec inhale 4 sec and exhale and 60-90 sec rest period (Kong et al., 2024).
5. Week 5 position (session duration 50min) from following positions:

   * Siting position (keeping the spine in upright and elongated position):

   Sitting position to train shoulder stabilizers with a coordinated interplay of the trunk and pelvic muscles. From this position, follow a manner of diaphragmatic breathing: 20 hyperventilation with 3 sec inhales ,6 sec exhales with 120-160 sec rest period .

   • Side Lying (Side Plank): Description: Participant lies on one side, supporting the body with the forearm and the lateral edge of the foot, while maintaining a neutral spine. The exercise focuses on activating the deep core musculature, including the obliques, transversus abdominis, and the lateral stabilizers of the pelvis and shoulder girdle. Participants are instructed to maintain optimal alignment of the head, spine, and pelvis while engaging in controlled diaphragmatic breathing.

   From this position, follow a breathing pattern aiming to train shoulder stabilizers with a coordinated interplay of the trunk and pelvic muscles. Diaphragmatic Breathing manner: 20 hyperventilation with 3 sec inhale, 6 sec exhale with 120-160 sec rest period.

   • Raising position (keep the spine forward and elongated and one leg kneeling): Description: Raising position with support on hands and feet. The hands are loaded equally on the thenar and hypothenar aspects, shoulders are aligned above the hands, feet are supported on the forefeet or on the entire soles, and the knees and hips are slightly flexed with the pelvis positioned higher than the head. The spine is elongated without any associated flexion or hyperextension.

   From this position, follow a manner of diaphragmatic breathing: 20 hyperventilation with 3 sec inhale ,6 sec exhale and 120-160 sec rest period .
6. Week 6 positions (session duration 55min) from following positions (Kong et al., 2024):

   • High Kneeling Position Keep the Spine Up Right and Elongated and One Leg Kneeling: High kneeling position maintaining shoulder stabilizers with a coordinated interplay of the trunk and pelvic muscles.

   From this position, follow a manner of diaphragmatic breathing: 20 hyperventilation with 3 sec inhale 6 sec and exhale and120-160 sec rest period (Kong et al., 2024).
   * Bear Position Description: Bear position with support on hands and feet, the hands are loaded equally on the thenar and hypothenar aspects, shoulders are aligned above the hands, feet are supported on forefeet or on the entire soles, and the knees and hips are slightly flexed with the pelvis positioned higher than the head, for training coordination of trunk and hip muscles.

   Order: Push the right hand and the left foot down to the floor and keep the spine as straight as possible at the same time. Do the same on the opposite side. Repeat a few times.

   From this position, follow a diaphragmatic breathing pattern keeping the spine elongated without any associated flexion or hyperextension: Diaphragmatic Breathing manner:20 hyperventilation with 3 sec inhales ,6 sec exhale with 120-160 sec rest period (Kong et al., 2024).

   • Squat Position: Description: Squat, with keeping the back straight, avoiding scapular retraction, forward drawn chest position, and anterior pelvic tilt, for training coordination of trunk and hip muscles.

   From this position, follow a manner of diaphragmatic breathing: 20 hyperventilation with 3 sec inhale, 6 sec exhale 120-160 sec rest period (Kong et al., 2024).

   • Standing Position (initial standing position) Description: Standing position, with the spine upright and the knees aligned above the big toes (the knee must not shift forward). Gradually, lower the hips to the level of the knees while keeping the arms relaxed at the side or reaching forward for training coordination of trunk and hip muscles. Gradually, lower the hips to the level of the knees while keeping the arms relaxed at the side or slightly reaching forward for training coordination of trunk and hip muscles.

   From this position, follow a manner of diaphragmatic breathing: 20 hyperventilation with 3 sec inhale 6 sec and exhale and 120-160 sec rest period (Kong et al., 2024).

   Statistical Analysis Statistical analysis was done by SPSS v26 (IBM Inc., Chicago, IL, USA). The Shapiro-Wilks test and histograms were used to evaluate the normality of the distribution of data. Quantitative parametric variables were presented as mean and standard deviation (SD) and compared between the two groups utilizing unpaired Student's T- test. Quantitative non-parametric data was presented as median and interquartile range (IQR) and was analyzed by Mann Whitney-test. Qualitative variables were presented as frequency and percentage (%) and were analyzed utilizing the Chi-square test or Fisher's exact test when appropriate. A two tailed P value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 34 years

Post-partum (3 to 6 months after delivery)

Diagnosed with mechanical low back pain

Body Mass Index (BMI) between 25 and 35 kg/m²

Medically stable and provided written informed consent

Exclusion Criteria:

Use of analgesics, anti-inflammatories, or any physical therapy interventions during the study period

History of severe trauma, skeletal injury, fracture, or neurological/chronic inflammatory disorders

Presence of malignancies (primary or metastatic) or osteoporosis

Diagnosed with chronic neuromuscular conditions

Failure to comply with instructions or attend regular sessions

-

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline (Week 0) and Post-Treatment (After 6 Weeks of Intervention)
  Assessed using the Numeric Pain Rating Scale (NPRS) - a subjective self-reported scale ranging from 0 (no pain) to 10 (worst imaginable pain).
Functional Disability | Baseline (Week 0) and Post-Treatment (After 6 Weeks of Intervention)
  Evaluated using the Modified Oswestry Disability Questionnaire (MODQ) - a validated tool for measuring limitations in daily activities due to low back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
This randomized controlled trial aimed to evaluate the effectiveness of Dynamic Neuromuscular Stabilization (DNS) in reducing pain and improving functional disability in women with post-partum low back pain (PLBP).
  A total of 60 post-partum women, aged 18-34 years, within 3 to 6 months post-delivery, and with BMI 25-35 kg/m², were randomly assigned to one of two groups:Intervention Group (n=30): Received conventional physiotherapy (ultrasound therapy and infrared therapy) combined with DNS exercises.
  Control Group (n=30): Received the same conventional physiotherapy without DNS.
  Both groups underwent three sessions per week for six weeks. Outcomes were assessed using the Numeric Pain Rating Scale (NPRS) and the Modified Oswestry Disability Questionnaire (MODQ) at baseline and after 6 weeks.
  The primary aim was to determine whether integrating DNS into standard physiotherapy results in superior outcom